CLINICAL TRIAL: NCT07292571
Title: SPECT/CT Imaging of Different Types of HER2 Expression in Breast Cancer Using Technetium-99m-labelled Affibody [99mTc]Tc -ZHER2:4107
Brief Title: Evaluation of Different Types of HER2 Expression in Breast Cancer Using [99mTc]Tc -ZHER2:4107
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HER2 expression level imaging
Record Dates: First submitted 2025-12-01; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Primary Breast Cancer
Keywords: [99mTc]Tc -ZHER2:4107; Breast Cancer; HER2 expression
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HER2-positive status (IHC 3+) (Experimental): Patients with HER2-positive status (IHC 3+)
  Interventions: Drug: Injection of [99mTc]Tc-ZHER2:4107, SPECT/CT
- IHC 1+ HER2 expression (Experimental): Patients with IHC 1+ HER2 expression
  Interventions: Drug: Injection of [99mTc]Tc-ZHER2:4107, SPECT/CT
- IHC 0 HER2 expression (Experimental): Patients with IHC 0 HER2 expression
  Interventions: Drug: Injection of [99mTc]Tc-ZHER2:4107, SPECT/CT

INTERVENTIONS:
Drug: Injection of [99mTc]Tc-ZHER2:4107, SPECT/CT — One single injection of [99mTc]Tc-ZHER2:4107, followed by SPECT/CT imaging 2 hours after injection
  Other Names: SPECT/CT Imaging Using Technetium-99m-labelled Affibody [99mTc]Tc -ZHER2:4107

SUMMARY:
The study should evaluate the [99mTc]Tc -ZHER2:4107 accumulation in primary tumour of breast cancer patients with different HER2 expression

DETAILED DESCRIPTION:
To determine different HER2 expression in primary breast cancer patients before any system or local treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years of age
2. Availability of results from HER2 status previously determined on material from the primary tumor and metastatic LN, either a. HER2-positive, defined as a DAKO HercepTest™ score of 3+ or FISH positive or b. HER2-negative, defined as a DAKO HercepTest™ score of 0 or 1+; or else if 2+ then FISH negative
3. Hematological, liver and renal function test results within the following limits:

   * White blood cell count: > 2.0 x 109/L
   * Hemoglobin: > 80 g/L
   * Platelets: > 50.0 x 109/L
   * ALT, ALP, AST: =< 5.0 times Upper Limit of Normal
   * Bilirubin =< 2.0 times Upper Limit of Normal
   * Serum creatinine: Within Normal Limits
4. A negative pregnancy test for all patients of childbearing potential. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception for at least 30 days after study termination
5. Subject is capable to undergo the diagnostic investigations to be performed in the study
6. Informed consent

Exclusion Criteria:

1. Any system therapy (chemo-/targeted therapy)
2. Second, non-breast malignancy
3. Active current autoimmune disease or history of autoimmune disease
4. Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening), known HIV positive or chronically active hepatitis B or C
5. Administration of other investigational medicinal product within 30 days of screening
6. Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with primary breast cancer
Enrollment: 50 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
[99mTc]Tc -ZHER2:4107 uptake in primary breast tumor | 2 hours
  SPECT/СT-based [99mTc]Tc -ZHER2:4107 uptake in primary breast tumor with different HER2 expression (SUVmax)
[99mTc]Tc -ZHER2:4107 background uptake | 2 hours
  SPECT-based [99mTc]Tc -ZHER2:41 background uptake value (SUVmax)
Tumor-to-background ratio | 2 hours
  The SPECT/CT-based tumor-to-background ratio will be calculated as follows: the value of [99mTc]Tc -ZHER2:41 uptake coinciding with tumor lesions (counts) will be divided by the value of [99mTc]Tc -ZHER2:41 uptake coinciding with the regions without pathological findings (SUVmax)

SECONDARY OUTCOMES:
Differentiation of HER2 expression in primary tumors | 2 hours
  To evaluate the threshold values of [99mTc]Tc -ZHER2:4107 accumulation for differentiation of HER2 expression in primary tumors in breast cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I Chernov, MD, Prof, Principal Investigator — Tomsk NRMC
Locations (1):
- Cancer Research Institute of Tomsk National Research Medical Center of the Russian Academy of Sciences, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Proposals may be submitted up to 36 months following publication of the results of the trial. After 36 months, the data will be available in the Center's data ware house but without investigator support other than deposited metadata.
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.